CLINICAL TRIAL: NCT03090373
Title: The Effect of Surface Acoustic Waves on the Prevention of Bacterial Colonization in Longterm Indwelling Urinary Catheters
Brief Title: The Effect of Surface Acoustic Waves on the Prevention of Colonization in Longterm Indwelling Urinary Caatheters
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rosenblum, Jonathan I., DPM (Individual)
Collaborators: Nanovibronix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: US-2
Record Dates: First submitted 2017-03-20; First posted 2017-03-24 (Actual); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Baacterial Colonization; Urinary Tract Infections
Keywords: Catheter; UTI's
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Intervention Model Description: This is a double blinded, randomized controlled trial. All involved will be blinded as to whether the supplied UroShield device is active or a sham.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The UroShield device actuator will activate and create the hum, which is the only sign of its working even in the active device. While the active device will transmit Surface Acoustic Waves, the sham device will work but will not transmit any acoustic waves.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Sham Comparator): At catheter replacement subjects will have a sham UroShield device attached to the external portion of the catheter and have it activated for 30 days.
  Standard of care for the upkeep and cleanliness of the catheter will be adhered to.
  At both the baseline and at the conclusion of 30 days, the distal end of the catheter will be collected as well as a sample of retained urine from the bladder and these samples will be evaluated for bacterial colonization.
  Interventions: Device: UroShield
- Treatment Group (Active Comparator): At catheter replacement subjects will have an active UroShield device attached to the external portion of the catheter and have it activated for 30 days.
  Standard of care for the upkeep and cleanliness of the catheter will be adhered to.
  At both the baseline and at the conclusion of 30 days, the distal end of the catheter will be collected as well as a sample of retained urine from the bladder and these samples will be evaluated for bacterial colonization.
  Interventions: Device: UroShield

INTERVENTIONS:
Device: UroShield — The UroShield is an externally applied acoustic actuator which generates surface acoustic waves and transmits them along the length of the catheter. The device does not come in direct contact with the subjects.
  Other Names: Surface Acoustic Wave Actuator

SUMMARY:
This is a double blinded rct to evaluate the effect of the UroShield SAW transducer on preventing bacterial colonization in longterm indwelling catheters. The duration of the trial is 30 days. The investigator will be quantifying the number of bacterial colonies in the urinary catheter and in the bladder in both the treatment and control group.

DETAILED DESCRIPTION:
This is a double blinded Randomized controoled trial of 30 days duration. The trial device is the Uroshield, SAW device which is an externally applied device attached to the external portion of the urinary catheter.

Subjects will be randomized to a control group and the treatment group. The control group will receive standard of care for the care of indwelling urinary catheters, while being attached to a sham UroShield device. The treatment group will receive the same standard of care treatment but will be attached to an active UroShield SAW device.

At baseline and again at 30 days, both the catheter and retained urine from the bladder will be evaluated for the number of live colonies. These numbers will be evaluated to see if there is a difference between the active and sham devices.

ELIGIBILITY:
Inclusion Criteria:

* Currently being treated with an indwelling urinary catheter for at least 30 days.
* Ability to sign informed consent or have someone authorized to sign informed consent.

Exclusion Criteria:

* Currently being treated for an active Urinary Tract infection.
* Previous treatment with Surface Acoustic Waves.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2018-03-01 (Estimated)

PRIMARY OUTCOMES:
Bacterial Colonization | 30 days
  Number of cultured colonies from both the Urinary Catheter and retained urine

CONTACTS AND LOCATIONS:
Locations (1):
- NanoVibronix, Elmsford, New York, United States

IPD SHARING:
Plan to Share IPD: No
Data will NOT be shared beyond the investigators of this study.